CLINICAL TRIAL: NCT05097703
Title: The Development and Pilot of a Sleep Resource for Carers of Pre-school Aged Children to be Used as Part of the Bedtime Routine
Brief Title: Sleep Resource for Carers of Pre-school Aged Children; a Development and Pilot Study
Acronym: SLEEPY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Surrey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FHMS 20-21 172 EGA
Record Dates: First submitted 2021-10-18; First posted 2021-10-28 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Sleep Hygiene
Keywords: Sleep intervention; Pre-school children; Caregivers
MeSH Terms: conditions — Sleep Hygiene

STUDY DESIGN:
Intervention Model Description: Participant randomly assigned to either an intervention arm or control arm. Intervention arm will receive the sleep resource and be asked to use it over a 4 week period where as the control group will not.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep Resource Intervention (Experimental): Half the participants in the study will be allocated to the intervention group. The resource will be sent to participants in this group, along with information about the research study and instructions for completing outcome measures. This will be followed up by a telephone call to ensure participants understand what is required of them and to answer any questions. All carers will be asked to complete questionnaires at baseline, immediately post intervention and at one-month post intervention; as well as sleep diaries for their child for the duration of the intervention period. Carers in the intervention group will also be asked to complete a diary of resource use as well as a feedback survey on their experience of using the resource.
  Carers in the intervention group will be asked that they use the resource with their child at bedtime for a minimum of three-days a week over a one-month period.
  Interventions: Behavioral: Sleep Resource
- Control (No Intervention): Participants randomised to the wait-list control group will be asked to complete pre, post and follow-up measures, as well as keep a sleep diary for the duration of the intervention period. They will then be sent the resource after the final outcome measures have been collected to use as they wish.

INTERVENTIONS:
Behavioral: Sleep Resource — The sleep resource is a card game to be played by children and caregivers as part of their bedtime routine. It includes exercises to help prepare the child for sleep, including deep breathing, mindfulness and light movement. Caregivers will be asked to use the resource for a minimum of three nights a week over a four week period, and complete pre and post outcome measures as well as sleep and resource use diaries for their children
  Arms: Sleep Resource Intervention

SUMMARY:
Evidence suggests sleep difficulties in pre-school children (aged 3-6 years) are highly prevalent and that carer knowledge of good sleep hygiene practices and the importance of them is relatively poor. Establishing a regular bedtime routine, involving activities shown to induce relaxation and prepare the child for sleep, is important in promoting optimal sleep duration and quality. However, there appears to be a lack of evidence-based resources that are empirically evaluated for carers to use with children within the family home. This study proposes to co-develop and pilot a new sleep resource. This will be an interactive storybook which guides children and their carers through a number of activities, designed to increase relaxation and prepare the child for sleep. A randomised control trial (RCT) design will be used, with an intervention group and a waitlist control group who will receive the resource at the end of the intervention period. Both groups will be asked to complete pre-intervention, post-intervention and follow-up measures; as well as keep sleep diaries for their children for the duration of the intervention period. The intervention group will also be asked to keep a diary of resource use and then to complete a feedback survey post-intervention. They will be asked to use the resource for a minimum of three days a week for a one-month period. This pilot aims to assess the acceptability of the resource and provide initial findings in terms of its efficacy on a range of sleep related outcomes.

DETAILED DESCRIPTION:
Typically, 3-6-year olds are estimated to require around 10-12 hours of sleep per day (The Sleep Council, 2019). This is thought to be essential for healthy growth and wellbeing, and is significantly associated with predictors of adult health (Bathory & Tomopoulos, 2017). Sleep disturbances and difficulties are found to be highly prevalent amongst infants and young children (Honaker & Meltzer, 2014). The literature estimates between 25% to 50% of pre-school aged children get too little sleep (Owens & Mindell, 2011), and a quarter of parents report sleep difficulties in their child's first five years of life (Bathory & Tomopoulos, 2017). This is a concern as evidence suggests early childhood to be a critical time for establishing sleep habits which have implications for sleep quality throughout the lifespan (Bonuck, Blank, True-Felt & Chervin, 2016). Research also shows a well-established link between sleep and long-term health outcomes for children. A recent review shows poor sleep to negatively effect physical health factors such as weight problems, as well as cognitive development, cognitive performance and behavioural functioning (Spruyt, 2019). Thinking more broadly about the impact on families, sleep problems in children have been found to impact the quality of maternal sleep, which then acts as a significant predictor of maternal mood, stress and fatigue (Meltzer & Mindell, 2007). Mindell and Williamson (2018) highlight that investing in not only interventions for disordered sleep but preventative strategies to promote healthy sleep is therefore essential in promoting positive health outcomes for children and their family systems.

Implementing sleep hygiene practices with children has been found to be positively associated with better sleep across a range of ages (Mindell, Meltzer, Carskadon & Chervin, 2009). Sleep hygiene can be defined as a set of specific behaviours and activities that are conducive to increasing healthy and adequate sleep (Perlis, Smith & Pigeon, 2005). This includes the consideration of factors such as environmental noise, bedroom environment, light exposure, exercise, temperature and electronic device use (Richdale & Schreck, 2019). Mindell and Williamson (2018) also suggest appropriate communication and contact with carer as an important aspect of sleep hygiene. The literature suggests that such techniques should be encompassed within a regular and structured bedtime routine to be most effective. Following a bedtime routine is associated with positive sleep outcomes; such as earlier bedtimes, increased sleep duration, reduced night time awakenings and reported caregiver sleep quality (Mindell and Williamson, 2018). Such outcomes have been observed in as little as two weeks from implementing sleep hygiene practices (Mindell, Leichman, Lee, Williamson & Walters, 2017). Encouraging bedtime routines that include sleep hygiene practices could therefore be a cost-effective way to promote positive childhood sleep outcomes, which could then have beneficial effects on a broad range of child development factors. Despite this, research suggests that caregiver knowledge in regards to their children's sleep habits is poor (McDowall, Galland, Campbell & Elder, 2017). Studies have shown increased knowledge of sleep hygiene to be associated with an increased number of positive sleep practices and increased sleep duration in young children (Owens & Jones, 2011). It has therefore been suggested that caregiver education on sleep hygiene could be used as a first line intervention for sleep problems in young children (McDowall, Galland, Campbell & Elder, 2017). This indicates that preventative interventions and resources for childhood sleep problems would likely benefit by including a degree of caregiver education.

Evidence-based interventions to promote healthy sleep habits in young children have largely focused on sub-groups of children and so may not be transferable to the general population (Busch, Altenburg, Harmsen and Chinapaw, 2017). For example, sleep interventions have been developed for children with autistic spectrum condition (Johnson et al., 2013; Turner & Johnson, 2013), intellectual disabilities (Stuttard, Beresford, Clarke, Beecham & Curtis, 2015), children with lymphoblastic leukaemia (Zupanec, Jones, McRae, Papaconstantinou, Weston & Stremler, 2017), those with specific sleep difficulties (Schlarb & Brandhorst, 2012; Kuhle, Urschitz, Eitner & Poets, 2009), as well as children living in socioeconomic adversity (Caldwell, Ordway, Sadler & Redeker, 2020; Ordway et al., 2020). In terms of interventions for the general population to promote healthy sleep, Busch, Altenburg, Harmsen and Chinapaw (2017) provide a review of those developed for children aged 4-12 years. They conclude that due to few high-quality studies, the effectiveness of any specific intervention strategy is inconclusive. They recommend the need for further evaluation of systematically developed interventions to encourage positive sleep habits in children. This current study's investigators argue the need for further research evidence examining which methods are effective in promoting healthy sleep in pre-school aged children, to then aid the development of widely accessible evidence-based resources.

Resources (e.g. storybooks, games) designed to be used with young children before bed are widely available. However, the efficacy of these in terms of promoting positive sleep outcomes relies mainly on anecdotal evidence from carer in the form of online reviews and blogs. Resources that have been evaluated in research for this age group tend to be in the form of educational interventions rather than ones that can be used at home. For example, the 'Sweet Dreamzzz Early Childhood Sleep Education program (Wilson, Miller, Bonuck, Lumeng & Chevrin, 2014) was developed for pre-school children and parents. This included a one-off workshop for parents and a two-week classroom curriculum for children to help establish bedtime routines involving positive sleep hygiene activities. Results included an increase of 30 minutes per night for children's sleep at one-month follow-up and increased parental knowledge of sleep hygiene practices; though this effect was not lasting. Schlarb and Branhorst (2012) developed an internet-based intervention, 'Mini-KiSS Online', for sleep disturbances in children aged 6-months to 4-years and their parents. Parents attended six online intervention sessions which included psychoeducation on sleep and implementing strategies to promote sleep hygiene including; imaginational exercises, bedtime stories, improving sleep environment; cognitive-behavioural techniques and relaxation exercises. Results indicate the intervention was highly accepted by parents and included improvements in falling asleep, less night time awakenings and less bedtime resistance. Though effect sizes were small to medium and results were limited by a high dropout rate (46%). Educational treatment programs rely on carer to independently implement learnt techniques which may be a reason for high dropout rates, as well as a high variation in how the strategies are implemented. This suggests that carer may benefit from resources they can use within the home, to help scaffold the bedtime routine and promote sleep hygiene activities in 'real time' with their children.

In terms of an evaluated resource that can be used at home, one study evaluated the game 'Perfect Bedroom: learn to sleep well'. This is a digital interactive game for 7-9-year olds, which encourages children to map out their bedtime routine to include sleep promoting activities and limit negative sleep hygiene activities such as the use of electronic devices. Preliminary results indicated the potential for this tool to be effective in promoting healthy sleep habits (Almondes & Leonardo, 2019), though the sample size was small (n=13). The authors also described this as the first study that used a 'serious game' (game designed for a primary purpose other than entertainment) to promote healthy sleep habits in children. In terms of study's evaluating serious games that promote healthy sleep habits for a younger age group in the home environment, this current project would therefore be the first to our knowledge to do so.

The literature highlights a need for the development and evaluation of evidence-based preventative resources that can be used at home as part of a child's bedtime routine. This study aims to provide a resource that pre-school children can play before bedtime with carers; in which they follow the characters on a journey through a fictional land, helping its inhabitants get a good night's sleep along the way. This will work by incorporating and encouraging positive sleep hygiene practices and relaxation exercises. It will include evidence-based practices shown to aid relaxation, using elements of mindfulness, deep breathing, imagery techniques and muscular relaxation. It will also include soothing activities and an appropriate level of child-caregiver interaction. The intervention is novel in that it aims to support children's sleep practices within the home environment, and therefore will have strong ecological validity. This research project therefore aims to develop and evaluate the sleep resource on a range of outcomes for both children and carer when played regularly together before bedtime.

ELIGIBILITY:
Inclusion Criteria:

* Carer-child dyads (3-6 years old) who feel their child could benefit from a resource designed to improve sleep outcomes.
* Fluent in English.
* Carers must hold legal parental responsibility for the child taking part in the study with them and be able to provide consent on their behalf.

Exclusion Criteria:

* Children who have a diagnosis of neurological disorder, cardiovascular or genetic diseases.
* Carers and or child unable to understand English.
* Carers who are not regularly available to assist children with the bedtime routine (e.g. do not live in the family home).

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2021-11-29 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Change in Carer reported child sleep diaries | 4 week period from baseline
  Carer to fill out sleep diary for child every day for four week period. To include time put to bed, time taken to fall asleep, frequency and duration of night time awakenings and time woke in morning.
Change in Resource use diaries | 4 week period from baseline
  Carer to fill out for child every day for four week period. To include time started using resource, length of time playing and the setting played in (e.g. bedroom, lounge).
Outcome of Feedback survey | 1 month
  Intervention group carers to complete feedback survey on the acceptability and utility of the resource. To include quantitative and qualitative feedback.

SECONDARY OUTCOMES:
Change in Children's Sleep-Wake Scale (CSWS) (LeBourgeois & Harsh, 2016) | Baseline, 1 month and 2 month post follow ups
  A caregiver report measure of behavioural sleep quality for 2 to 8 year old children. It quantitatively assesses 5 distinct behavioural dimensions of sleep quality, including Going to Bed, Falling Asleep, Maintaining Sleep, Reinitiating Sleep, and Returning to Wakefulness.
Change in General Sleep Information (GSI) (Akacem, Wright & LeBourgeois, 2016) | Baseline, 1 month and 2 month post follow ups
  A caregiver report form for 2 to 12 year old children. Assess bed time routine and timings, night time awakenings and parent view of child sleep quality and function.
Change in Strengths and Difficulties Questionnaire, parent version (SDQ) (Goodman, 1997) | Baseline, 1 month and 2 month post follow ups
  A brief behavioural screening guide for 3 to 16 year olds. It includes 25 questions on psychological attributes.
Change in Parenting Stress Scale (PSS) (Berry & Jones, 1995) | Baseline, 1 month and 2 month post follow ups
  An 18 item questionnaire assessing parents' views of their parenting role, exploring both positive and negative aspects of parenthood.
Change in Parent-Child Sleep Interactions Scale (PCSIS) (Alfano, Smith, Reynolds, Reddy & Dougherty, 2013) | Baseline, 1 month and 2 month post follow ups
  A caregiver report measure designed to assess a wide range of bedtime behaviours.

OTHER OUTCOMES:
Demographics | Baseline
  Household characteristics

CONTACTS AND LOCATIONS:
Overall Officials: Alex J Tapping, BSc MSc, Principal Investigator — University of Surrey
Locations (1):
- Alex Tapping, Guildford, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alfano CA, Smith VC, Reynolds KC, Reddy R, Dougherty LR. The Parent-Child Sleep Interactions Scale (PSIS) for preschoolers: factor structure and initial psychometric properties. J Clin Sleep Med. 2013 Nov 15;9(11):1153-60. doi: 10.5664/jcsm.3156. PMID 24235896
- [Background] Almondes KM, Leonardo MEM. Games as education tools. Sleep Sci. 2019 Apr-Jun;12(2):100-105. doi: 10.5935/1984-0063.20190069. PMID 31879542
- [Background] Bathory E, Tomopoulos S. Sleep Regulation, Physiology and Development, Sleep Duration and Patterns, and Sleep Hygiene in Infants, Toddlers, and Preschool-Age Children. Curr Probl Pediatr Adolesc Health Care. 2017 Feb;47(2):29-42. doi: 10.1016/j.cppeds.2016.12.001. Epub 2017 Jan 20. PMID 28117135
- [Background] Berry, J. O., & Jones, W. H. (1995). The Parental Stress Scale: Initial psychometric evidence. Journal of Social and Personal Relationships, 12(3), 463-472
- [Background] Bonuck KA, Blank A, True-Felt B, Chervin R. Promoting Sleep Health Among Families of Young Children in Head Start: Protocol for a Social-Ecological Approach. Prev Chronic Dis. 2016 Sep 1;13:E121. doi: 10.5888/pcd13.160144. PMID 27584877
- [Background] Busch V, Altenburg TM, Harmsen IA, Chinapaw MJ. Interventions that stimulate healthy sleep in school-aged children: a systematic literature review. Eur J Public Health. 2017 Feb 1;27(1):53-65. doi: 10.1093/eurpub/ckw140. PMID 28177474
- [Background] Caldwell BA, Ordway MR, Sadler LS, Redeker NS. Parent Perspectives on Sleep and Sleep Habits Among Young Children Living With Economic Adversity. J Pediatr Health Care. 2020 Jan-Feb;34(1):10-22. doi: 10.1016/j.pedhc.2019.06.006. Epub 2019 Aug 31. PMID 31477491
- [Background] Goodman R. The Strengths and Difficulties Questionnaire: a research note. J Child Psychol Psychiatry. 1997 Jul;38(5):581-6. doi: 10.1111/j.1469-7610.1997.tb01545.x. PMID 9255702
- [Background] Honaker SM, Meltzer LJ. Bedtime problems and night wakings in young children: an update of the evidence. Paediatr Respir Rev. 2014 Dec;15(4):333-9. doi: 10.1016/j.prrv.2014.04.011. Epub 2014 Apr 13. PMID 24908611
- [Background] Johnson CR, Turner KS, Foldes E, Brooks MM, Kronk R, Wiggs L. Behavioral parent training to address sleep disturbances in young children with autism spectrum disorder: a pilot trial. Sleep Med. 2013 Oct;14(10):995-1004. doi: 10.1016/j.sleep.2013.05.013. Epub 2013 Aug 27. PMID 23993773
- [Background] Kuhle S, Urschitz MS, Eitner S, Poets CF. Interventions for obstructive sleep apnea in children: a systematic review. Sleep Med Rev. 2009 Apr;13(2):123-31. doi: 10.1016/j.smrv.2008.07.006. Epub 2008 Dec 6. PMID 19059794
- [Background] LeBourgeois MK, Harsh JR. Development and psychometric evaluation of the Children's Sleep-Wake Scale<sup/> Sleep Health. 2016 Sep;2(3):198-204. doi: 10.1016/j.sleh.2016.04.001. PMID 28066802
- [Background] McDowall PS, Galland BC, Campbell AJ, Elder DE. Parent knowledge of children's sleep: A systematic review. Sleep Med Rev. 2017 Feb;31:39-47. doi: 10.1016/j.smrv.2016.01.002. Epub 2016 Jan 14. PMID 26899741
- [Background] Meltzer LJ, Mindell JA. Relationship between child sleep disturbances and maternal sleep, mood, and parenting stress: a pilot study. J Fam Psychol. 2007 Mar;21(1):67-73. doi: 10.1037/0893-3200.21.1.67. PMID 17371111
- [Background] Mindell JA, Leichman ES, Lee C, Williamson AA, Walters RM. Implementation of a nightly bedtime routine: How quickly do things improve? Infant Behav Dev. 2017 Nov;49:220-227. doi: 10.1016/j.infbeh.2017.09.013. Epub 2017 Oct 3. PMID 28985580
- [Background] Mindell JA, Meltzer LJ, Carskadon MA, Chervin RD. Developmental aspects of sleep hygiene: findings from the 2004 National Sleep Foundation Sleep in America Poll. Sleep Med. 2009 Aug;10(7):771-9. doi: 10.1016/j.sleep.2008.07.016. Epub 2009 Mar 12. PMID 19285450
- [Background] Mindell JA, Williamson AA. Benefits of a bedtime routine in young children: Sleep, development, and beyond. Sleep Med Rev. 2018 Aug;40:93-108. doi: 10.1016/j.smrv.2017.10.007. Epub 2017 Nov 6. PMID 29195725
- [Background] Perlis, M. L., Smith, M. T., & Pigeon, W. R. (2005). Etiology and pathophysiology of insomnia. Principles and practice of sleep medicine, 4, 714-725.
- [Background] Ordway MR, Sadler LS, Jeon S, O'Connell M, Banasiak N, Fenick AM, Crowley AA, Canapari C, Redeker NS. Sleep health in young children living with socioeconomic adversity. Res Nurs Health. 2020 Aug;43(4):329-340. doi: 10.1002/nur.22023. Epub 2020 Apr 19. PMID 32306413
- [Background] Owens JA, Jones C. Parental knowledge of healthy sleep in young children: results of a primary care clinic survey. J Dev Behav Pediatr. 2011 Jul-Aug;32(6):447-53. doi: 10.1097/DBP.0b013e31821bd20b. PMID 21546852
- [Background] Owens JA, Mindell JA. Pediatric insomnia. Pediatr Clin North Am. 2011 Jun;58(3):555-69. doi: 10.1016/j.pcl.2011.03.011. PMID 21600342
- [Background] Richdale, A. L., & Schreck, K. A. (2019). Examining sleep hygiene factors and sleep in young children with and without autism spectrum disorder. Research in Autism Spectrum Disorders, 57, 154-162.
- [Background] Schlarb AA, Brandhorst I. Mini-KiSS Online: an Internet-based intervention program for parents of young children with sleep problems - influence on parental behavior and children's sleep. Nat Sci Sleep. 2012 Mar 12;4:41-52. doi: 10.2147/NSS.S28337. Print 2012. PMID 23620677
- [Background] Spruyt K. A review of developmental consequences of poor sleep in childhood. Sleep Med. 2019 Aug;60:3-12. doi: 10.1016/j.sleep.2018.11.021. Epub 2018 Dec 15. PMID 30660750
- [Background] Stuttard L, Beresford B, Clarke S, Beecham J, Curtis J. A preliminary investigation into the effectiveness of a group-delivered sleep management intervention for parents of children with intellectual disabilities. J Intellect Disabil. 2015 Dec;19(4):342-55. doi: 10.1177/1744629515576610. Epub 2015 Mar 19. PMID 25792540
- [Background] Turner, K. S., & Johnson, C. R. (2013). Behavioral interventions to address sleep disturbances in children with autism spectrum disorders: a review. Topics in Early Childhood Special Education, 33(3), 144-152.
- [Background] Wilson KE, Miller AL, Bonuck K, Lumeng JC, Chervin RD. Evaluation of a sleep education program for low-income preschool children and their families. Sleep. 2014 Jun 1;37(6):1117-25. doi: 10.5665/sleep.3774. PMID 24882907
- [Background] Zupanec S, Jones H, McRae L, Papaconstantinou E, Weston J, Stremler R. A Sleep Hygiene and Relaxation Intervention for Children With Acute Lymphoblastic Leukemia: A Pilot Randomized Controlled Trial. Cancer Nurs. 2017 Nov/Dec;40(6):488-496. doi: 10.1097/NCC.0000000000000457. PMID 27922922
- See also: Sleep Council recommendations — http://sleepcouncil.org.uk/how-much-sleep-does-my-child-need/